CLINICAL TRIAL: NCT05759949
Title: A First-in-Human Study of PI3Kα Inhibitor, RLY-5836, in Combination With Targeted and Endocrine Therapies in Participants With Advanced Breast Cancer and as a Single Agent in Advanced Solid Tumors
Brief Title: First-in-Human Study of RLY-5836 in Advanced Breast Cancer and Other Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Relay Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RLY-5836-101
Record Dates: First submitted 2023-01-23; First posted 2023-03-08 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: PIK3CA Mutation; Solid Tumor, Adult; HER2-negative Breast Cancer; Breast Cancer; Metastatic Breast Cancer; Advanced Breast Cancer; Unresectable Solid Tumor; Hormone Receptor Positive Tumor
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; palbociclib; ribociclib; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- RLY-5836 Single Agent Arm (Experimental): RLY-5836 single agent arm for participants with unresectable or metastatic solid tumors
  Interventions: Drug: RLY-5836
- RLY-5836 + Fulvestrant Arm (Experimental): RLY-5836 + fulvestrant combination arm for participants with HR+, HER2- locally advanced or metastatic breast cancer
  Interventions: Drug: RLY-5836; Drug: Fulvestrant
- RLY-5836 + Palbociclib + Fulvestrant Arm (Experimental): RLY-5836 + palbociclib + fulvestrant triple combination arm for participants with HR+, HER2- locally advanced or metastatic breast cancer
  Interventions: Drug: RLY-5836; Drug: Fulvestrant; Drug: Palbociclib
- RLY-5836 + Ribociclib + Fulvestrant Arm (Experimental): RLY-5836 + ribociclib + fulvestrant triple combination arm for participants with HR+, HER2- locally advanced or metastatic breast cancer
  Interventions: Drug: RLY-5836; Drug: Fulvestrant; Drug: Ribociclib
- RLY-5836 + Abemaciclib + Fulvestrant Arm (Experimental): RLY-5836 + abemaciclib + fulvestrant triple combination arm for participants with HR+, HER2- locally advanced or metastatic breast cancer
  Interventions: Drug: RLY-5836; Drug: Fulvestrant; Drug: Abemaciclib

INTERVENTIONS:
Drug: RLY-5836 — RLY-5836 is a mutant-selective, oral PI3Kα inhibitor.
Drug: Fulvestrant — Fulvestrant (500 mg) is administered IM into the buttocks (gluteal area) slowly (1 to 2 minutes per injection) as 2×5 mL injections, 1 in each buttock, on Cycle 1 Day 1, Cycle 1 Day 15, and Day 1 of each subsequent cycle.
  Other Names: Faslodex
  Arms: RLY-5836 + Abemaciclib + Fulvestrant Arm; RLY-5836 + Fulvestrant Arm; RLY-5836 + Palbociclib + Fulvestrant Arm; RLY-5836 + Ribociclib + Fulvestrant Arm
Drug: Palbociclib — Palbociclib 125 mg once daily is taken orally in combination with RLY-5836 and fulvestrant for 28-day cycles that include 21 days of treatment followed by 7 days off treatment.
  Other Names: Ibrance
  Arms: RLY-5836 + Palbociclib + Fulvestrant Arm
Drug: Ribociclib — Ribociclib 600 mg once daily is taken orally in combination with RLY-5836 and fulvestrant for 28-day cycles that include 21 days of treatment followed by 7 days off treatment.
  Other Names: Kisqali
  Arms: RLY-5836 + Ribociclib + Fulvestrant Arm
Drug: Abemaciclib — Abemaciclib 150 mg BID will be taken orally in combination with RLY-5836 and fulvestrant for 28-day cycles.
  Other Names: Verzenio
  Arms: RLY-5836 + Abemaciclib + Fulvestrant Arm

SUMMARY:
This is a Phase 1, first-in-human, open-label study designed to evaluate the maximum tolerated dose (MTD), recommended phase 2 dose (RP2D), safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary anti-tumor activity of RLY-5836 in advanced solid tumors in participants harboring a PIK3CA mutation in blood and/or tumor per local assessment. The study consists of 2 parts, a dose escalation (Part 1) and a dose expansion (Part 2).

ELIGIBILITY:
Inclusion Criteria:

Patient has ECOG performance status of 0-1

One or more documented primary oncogenic PIK3CA mutation(s) in blood and/or tumor per local assessment

RLY-5836 single agent arm key inclusion criteria

* Disease that is refractory to standard therapy, intolerant to standard therapy, or participant has declined standard therapy.
* A histologically or cytologically confirmed diagnosis of unresectable or metastatic solid tumor

Combination arms key inclusion criteria

* Males, postmenopausal females, or pre-/perimenopausal females previously treated with gonadotropin-releasing GnRH agonist at least 4 weeks prior to start of study drug with histologically or cytologically confirmed diagnosis of HR+, HER2- unresectable or metastatic breast cancer that is not amenable to curative therapy.
* Had previous treatment for advanced or metastatic breast cancer with antiestrogen therapy including, but not limited to, selective estrogen receptor degraders (e.g., fulvestrant), selective estrogen receptor modulators (e.g., tamoxifen), and aromatase inhibitors (AI) (letrozole, anastrozole, exemestane)
* Part 1: Prior PI3Kα inhibitor treatment is allowed if taken for < 14 days and not discontinued due to disease progression, hypersensitivity, or ≥ Grade 3 TEAEs.

Exclusion Criteria:

* Part 2: Prior treatment with PI3Kα inhibitors.
* Type 1 or Type 2 diabetes requiring antihyperglycemic medication, or fasting plasma glucose ≥140 mg/dL and glycosylated hemoglobin (HbA1c) ≥7.0%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of RLY-5836 | Cycle 1 (4-week cycle) of treatment for MTD and at the end of every cycle (4-week cycles) for RP2D until study discontinuation, approximately 24 months
Number of participants with any dose-limiting toxicity (DLT) | Cycle 1, up to 28 days.
Number of participants with adverse events (AEs) | Every cycle (4-week cycles) until study discontinuation, approximately 24 months
Number of participants with serious adverse events (SAEs) | Every cycle (4-week cycles) until study discontinuation, approximately 24 months

SECONDARY OUTCOMES:
PIK3CA genotype in blood and tumor tissue by next generation nucleic acid sequencing | Every cycle (4-week cycles) through Cycle 3 and every other cycle thereafter until study discontinuation, approximately 24 months
PK of RLY-5836: area under the concentration-time curve (AUC) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through end of treatment (4-week cycles), approximately 24 months
PK of RLY-5836: maximum plasma concentration (Cmax) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through end of treatment (4-week cycles), approximately 24 months
PK of RLY-5836: time to maximum concentration (tmax) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through end of treatment (4-week cycles), approximately 24 months
PK of RLY-5836: half-life (t½) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through end of treatment (4-week cycles), approximately 24 months
PK of RLY-5836: clearance following oral dose (CL/F) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through end of treatment (4-week cycles), approximately 24 months
Changes in circulating markers of glucose metabolism: changes in circulating glucose | Approximately every week in Cycle 1 (4-week cycle), every 2 weeks in Cycle 2 (4-week cycle), and every cycle through end of treatment (4-week cycles), approximately 24 months
Changes in circulating markers of glucose metabolism: changes in circulating insulin | Approximately every week in Cycle 1 (4-week cycle), every 2 weeks in Cycle 2 (4-week cycle), and every cycle through end of treatment (4-week cycles), approximately 24 months
Changes in circulating markers of glucose metabolism: changes in circulating C-peptide | Approximately every week in Cycle 1 (4-week cycle), every 2 weeks in Cycle 2 (4-week cycle), and every cycle through end of treatment (4-week cycles), approximately 24 months
Changes in circulating markers of glucose metabolism: changes in circulating glycosylated hemoglobin [HbA1c] | Approximately every week in Cycle 1 (4-week cycle), every 2 weeks in Cycle 2 (4-week cycle), and every cycle through end of treatment (4-week cycles), approximately 24 months
Preliminary antitumor activity of RLY-5836: duration of response (DOR) per Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) | Approximately every 8 weeks until progressive disease, approximately 36 months
Preliminary antitumor activity of RLY-5836: disease control rate (DCR) per Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) | Approximately every 8 weeks until progressive disease, approximately 36 months
Preliminary antitumor activity of RLY-5836: objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) | Approximately every 8 weeks until progressive disease, approximately 36 months

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - Community Cancer Center North, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center-Main Campus, New York, New York
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No